CLINICAL TRIAL: NCT06886399
Title: INVESTIGATION of the EFFICACY and SAFETY of the DRUG "AS-PROBIONORM" with the PARTICIPATION of PATIENTS with DYSBIOSIS (phase 2)
Brief Title: INVESTIGATION of the EFFICACY and SAFETY of the DRUG "AS-PROBIONORM"
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Industrial Microbiology LLP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ПМ-003-23г
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Intestinal Infections; Dysbacteriosis
Keywords: probiotic; intestinal infections; dysbiosis; lactic acid bacteria; phase 2 of clinical trial
MeSH Terms: conditions — Dysbiosis

STUDY DESIGN:
Intervention Model Description: Phase II of the clinical trial of the medicine included 210 study subjects with identified clinical and/or microbiological signs of dysbiosis. 3 groups of 70 research subjects will be formed.
  Group 1 - study subjects with an identified decrease in intestinal microflora activity; Group 2 - study subjects with an identified fungal (candidiasis) infection; Group 3 - study subjects with active pathogenic microflora.
  Study design: open-label, single-center, phase II of clinical trial. Dosage regimen for first group - 1 sachet (1 g) 2 times a day (morning and evening) 15 min prior food , with an interval of 12 hours. The total duration of study subjects' participation in the study is 28 days. Dosage regimen for the second and third groups - 2 sachet (2 g) 2 times a day (morning and evening) 15 min prior food , with an interval of 12 hours. The total duration of study subjects' participation in the study is 28 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects with identified clinical and/or microbiological signs of dysbiosis (Experimental): Dosage regimen for first group - 1 sachet (1 g) 2 times a day (morning and evening) 15 min prior food , with an interval of 12 hours. The total duration of study subjects' participation in the study is 28 days. Dosage regimen for the second and third groups - 2 sachet (2 g) 2 times a day (morning and evening) 15 min prior food , with an interval of 12 hours. The total duration of study subjects' participation in the study is 28 days.
  Interventions: Drug: "AS-Probionorm"

INTERVENTIONS:
Drug: "AS-Probionorm" — Phase II of the clinical trial of the medicine included 210 study subjects with identified clinical and/or microbiological signs of dysbiosis. 3 groups of 70 research subjects will be formed.
  Group 1 - study subjects with an identified decrease in intestinal microflora activity; Group 2 - study subjects with an identified fungal (candidiasis) infection; Group 3 - study subjects with active pathogenic microflora.
  Dosage regimen for first group - 1 sachet (1 g) 2 times a day (morning and evening) 15 min prior food , with an interval of 12 hours. The total duration of study subjects' participation in the study is 28 days. Dosage regimen for the second and third groups - 2 sachet (2 g) 2 times a day (morning and evening) 15 min prior food , with an interval of 12 hours. The total duration of study subjects' participation in the study is 28 days.

SUMMARY:
The subject of this clinical trial is the medicine "AS-Probionorm". Pharmacological group - Antidiarrheal drugs. Antidiarrheal microorganisms. Microorganisms that produce lactic acid.

The investigational probiotic medicine "AS-Probionorm" was created on the basis of an association of lactic acid bacteria with targeted action for oral use for the treatment of inflammatory and infectious diseases of the human gastrointestinal tract.

The second phase of a clinical trial is the study of a medicine conducted on volunteers to establish efficacy and safety.

According to this study, the aim of this clinical trial is to investigate the efficacy, safety, and optimal dosage regimen for the investigational medicinal product AS-Probionorm (powder in sachets of 1 gram) for oral administration in patients with dysbiosis.

Phase II of the clinical trial of the medicine included 210 study subjects with identified clinical and/or microbiological signs of dysbiosis. 3 groups of 70 research subjects will be formed.

Selection and Exclusion of Subjects: Prior to inclusion in a clinical trial, each trial subject must first sign an Informed Consent Form for Participation in the Study, followed by a screening examination of each subject, including a variety of procedures, medical history, and physical examination. Each subject participating in the survey will be assigned an identification number.

Study design: open-label, single-center, phase II of clinical trial. Dosage regimen for first group - 1 sachet (1 g) 2 times a day (morning and evening) 15 min prior food , with an interval of 12 hours. The total duration of study subjects' participation in the study is 28 days. Dosage regimen for the second and third groups - 2 sachet (2 g) 2 times a day (morning and evening) 15 min prior food , with an interval of 12 hours. The total duration of study subjects' participation in the study is 28 days.

Safety of the study drug: The safety assessment of AS-Probinorm (powder in sachets) is based on the results of dynamic monitoring of study subjects after they take the study drug for one day and for the next 42 days. The following data are used as the basis for the assessment: complaints, physical examination results, and results of laboratory and instrumental research methods.

The effectiveness of the drug will be evaluated based on the subjective experiences and sensations reported by patients, as well as objective data collected by the researchers during the study.

The degree of effectiveness of the studied drug will be assessed based on three categories:

* Intolerance - the appearance of local symptoms of allergy/pseudoallergy and systemic symptoms such as tachycardia (heart rate greater than 90 beats per minute for more than 30 minutes after administration), lowered blood pressure (lower than 100/60 mm Hg within 30 minutes of application), and serious adverse reactions.
* No adverse reactions
* Undesirable effects that are not considered serious Ethical and Legal Issues in Clinical Research: This clinical trial will be conducted in accordance with the principles set forth by the 18th World Medical Assembly (Helsinki, 1964) and the ICH guidelines for good clinical practice (GCP), and in accordance with all international and national laws and regulations.

DETAILED DESCRIPTION:
Dosage form of the medicine "AS-Probionorm" (powder for the preparation of solution for oral administration) - 1 g in a sachet for patients with dysbiosis.

Pharmacological group - Antidiarrheal drugs. Antidiarrheal microorganisms. Microorganisms that produce lactic acid.

Introduction:

Acute intestinal infections (AKI) are a significant health problem in all countries, including Kazakhstan. Due to their widespread prevalence, high incidence of moderate and severe forms, and potential complications, it is essential to find ways to improve treatment strategies for this group of illnesses.

Probiotics based on beneficial microorganisms from the gastrointestinal tract are increasingly being recommended for the treatment of intestinal and urinary tract infections instead of antibiotics worldwide. Lactic acid bacteria and bifidobacteria are among the most commonly used, as experts consider their pathogenic potential to be sufficiently low for oral administration at conventional doses. These medications quickly suppress harmful microbes and activate the immune system. Therefore, the modern strategy for the treatment of acute intestinal infections gives priority to therapeutic measures aimed at correcting intestinal microbiocenosis to eliminate the source of infection localized in the intestine.

The main idea is to conduct clinical studies of the domestic medicinal probiotic medicine "AS-Probionorm" based on the association of lactic acid bacteria of targeted action for oral use for the treatment of inflammatory and infectious diseases of the human gastrointestinal tract.

During the first phase of clinical trials, the investigational drug AS-Probionorm was found to be well tolerated, safe, and does not cause any undesirable side effects or dysbiotic disorders. It also does not cause allergic reactions, changes in blood formulas, levels of aminotransferases (ALT and AST), serum albumin, or blood sugar.

According to this study, the aim of this clinical trial is to investigate the efficacy, safety, and optimal dosage regimen for the investigational medicinal product AS-Probionorm (powder in sachets of 1 gram) for oral administration in patients with dysbiosis.

Phase II of the clinical trial of the medicine included 210 study subjects with identified clinical and/or microbiological signs of dysbiosis. 3 groups of 70 research subjects will be formed.

Group 1 - study subjects with an identified decrease in intestinal microflora activity; Group 2 - study subjects with an identified fungal (candidiasis) infection; Group 3 - study subjects with active pathogenic microflora.

Selection and Exclusion of Subjects: Prior to inclusion in a clinical trial, each trial subject must first sign an Informed Consent Form for Participation in the Study, followed by a screening examination of each subject, including a variety of procedures, medical history, and physical examination. Each subject participating in the survey will be assigned an identification number.

Study design: open-label, single-center, phase II of clinical trial. Dosage regimen for first group - 1 sachet (1 g) 2 times a day (morning and evening) 15 min prior food , with an interval of 12 hours. The total duration of study subjects' participation in the study is 28 days. Dosage regimen for the second and third groups - 2 sachet (2 g) 2 times a day (morning and evening) 15 min prior food , with an interval of 12 hours. The total duration of study subjects' participation in the study is 28 days.

To obtain information about the efficacy and safety of the investigational drug, the study subjects will be monitored for 42 days. The study will be performed on an outpatient basis. The total duration of the study subjects' participation in the study is 42 days. On days 1, 14, 28, 42, medical examinations and laboratory tests will be conducted.

Safety of the study drug: The safety assessment of AS-Probinorm (powder in sachets) is based on the results of dynamic monitoring of study subjects after they take the study drug for one day and for the next 42 days. The following data are used as the basis for the assessment: complaints, physical examination results, and results of laboratory and instrumental research methods.

Safety assessment criteria: absence of dysbiotic disorders, absence of allergic manifestations, absence of clinically significant changes in the blood formula, determination of the level of aminotransferases (ALT, AST), serum albumin, sugar, blood bilirubin, reactions from the gastrointestinal tract, general somatic state (body temperature, blood pressure, heart rate) of the study subjects during research. Absence of undesirable reactions. At the recommended doses, the investigational drug does not cause a negative reaction of the body.

The effectiveness of the drug will be evaluated based on the subjective experiences and sensations reported by patients, as well as objective data collected by the researchers during the study.

The degree of effectiveness of the studied drug will be assessed based on three categories:

* Intolerance - the appearance of local symptoms of allergy/pseudoallergy and systemic symptoms such as tachycardia (heart rate greater than 90 beats per minute for more than 30 minutes after administration), lowered blood pressure (lower than 100/60 mm Hg within 30 minutes of application), and serious adverse reactions.
* No adverse reactions
* Undesirable effects that are not considered serious Ethical and Legal Issues in Clinical Research: This clinical trial will be conducted in accordance with the principles set forth by the 18th World Medical Assembly (Helsinki, 1964) and the ICH guidelines for good clinical practice (GCP), and in accordance with all international and national laws and regulations.

Data analysis was carried out using several statistical methods: Student's t-test (Student's t-test), parametric and Met: U-test of what-Whitney (Mann Whitney U test), Kruskal Wallis test (Kruskal Wallis test H), Chi-square criterion (Chi-squared test).

Data collection, maintenance and storage of records. Data collection will be carried out electronically and, partially, in paper form.

The Investigator must maintain all research documentation (electronic and paper) in confidence and take steps to prevent accidental or premature destruction of this documentation.

The Investigator must retain all study documentation for a minimum of fifteen (15) years after completion or premature termination of the clinical trial.

However, if a longer period is required, applicable legal requirements must be taken into account.

The investigator must notify the sponsor before destroying any important study documents following completion or premature termination of a clinical trial.

Financing and insurance. All financing and insurance issues will be determined in the agreement concluded between the Sponsor and the Contractor.

Publications. The Investigator agrees not to publish or report the study and/or its results without the prior written permission of the study sponsor, noting that the sponsor will not withhold such permission without reasonable cause. The researcher will not use the sponsor's name in any promotional material or publication without the sponsor's prior written consent. The sponsor will not use the name of the investigator and/or his/her collaborators in promotional materials or publications without first obtaining his/their written consent. The sponsor has the right to publish the study results at any time.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dysbiosis - Bacterial overgrowth syndrome (ICD-10 PK K63.8 Other specified intestinal diseases) of both sexes aged 18-50 years
* Patients with Irritable Bowel Syndrome (ICD-10 RC K58)
* Patients with Irritable bowel syndrome with diarrhea (ICD-10 RC K58.0)
* Patients with Irritable bowel syndrome without diarrhea (ICD-10 RC K58.9)
* Patients with verified health status, absence of chronic and acute systemic diseases and intestinal;
* For women, a negative pregnancy test and consent to adhere to adequate methods of contraception.
* A voluntary desire to participate in the study.

Exclusion Criteria:

* Subjects with a history of allergy to milk, and during screening (drug, pollen, and other types), individual hypersensitivity to the components of the drug;
* Subjects with chronic diseases (tuberculosis, hepatitis, HIV infection, diabetes mellitus, cancer, blood diseases), chronic renal failure, chronic liver failure, exacerbations of chronic diseases;
* Subjects who participate in parallel clinical trials of other medicines, or who have participated in them for 3 months. from the beginning of the current study;
* Subjects planning to participate in the research should not take any other medications for 2 weeks before the clinical trials of the test drug.;
* Subjects from the category of "vulnerable" (homeless, military personnel, the incapacitated, patients in urgent conditions, other persons who may be under pressure);
* Pregnancy and breast - feeding;
* The subject of the study does not agree to perform the procedures required by the protocol and is unable to adhere to the schedule of procedures.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-08-11 (Actual); Study Completion 2024-08-11 (Actual)

PRIMARY OUTCOMES:
Safety of the study drug: | 1 day of taking the drug for the next 42 days
  Safety of the study drug: The safety assessment of AS-Probinorm (powder in sachets) is based on the results of dynamic monitoring of study subjects after they take the study drug for one day and for the next 42 days. The following data are used as the basis for the assessment: complaints, physical examination results, and results of laboratory and instrumental research methods.
  Safety assessment criteria: absence of dysbiotic disorders, absence of allergic manifestations, absence of clinically significant changes in the blood formula, determination of the level of aminotransferases (ALT, AST), serum albumin, sugar, blood bilirubin, reactions from the gastrointestinal tract, general somatic state (body temperature, blood pressure, heart rate) of the study subjects during research. Absence of undesirable reactions. At the recommended doses, the investigational drug does not cause a negative reaction of the body.
The effectiveness of the drug | During 24 hours
  The effectiveness of the drug will be evaluated based on the subjective experiences and sensations reported by patients, as well as objective data collected by the researchers during the study.
  The degree of effectiveness of the studied drug will be assessed based on three categories:
  * Intolerance - the appearance of local symptoms of allergy/pseudoallergy and systemic symptoms such as tachycardia (heart rate greater than 90 beats per minute for more than 30 minutes after administration), lowered blood pressure (lower than 100/60 mm Hg within 30 minutes of application), and serious adverse reactions.
  * No adverse reactions
  * Undesirable effects that are not considered serious

CONTACTS AND LOCATIONS:
Overall Officials: Ilyas Kulmagambetov, Doctor of Med. Sc., Principal Investigator — Centre for Clinical Medicine and Research LLP
Locations (1):
- MIPO Clinic LLP, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1) A.K. Sadanov, N.N. Gavrilova, I.A. Ratnikova, S.E. Orazymbet, E.Zh. Shorabayev, Zh.T. Musabekov, R.Zh. Kaptagay, L.E. Protasyuk, L.A. Kosheleva, S.B. Dzhailyauova Association of bacteria for the production of a medicinal probiotic preparation with a wide spectrum of antimicrobial action // Microbiology and virology. - ISSN 2304-585X. - No. 1 (40) 2023. -- pp. 116-126.